CLINICAL TRIAL: NCT01818895
Title: Terminal Weaning of Mechanical Ventilation or Extubation in Anticipation of Death in the Intensive Care Unit: Impact on Relatives, Care Givers and the Dying Process - A Prospective, Multicenter, Observational Study
Brief Title: Terminal Weaning of Mechanical Ventilation or Extubation in Anticipation of Death in the Intensive Care Unit
Acronym: ARREVE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Collaborators: Poitiers University Hospital (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: CHD 018-13
Record Dates: First submitted 2013-03-21; First posted 2013-03-27 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Withdrawal; Anxiety; Depression; Posttraumatic Stress Disorder
Keywords: Mechanical ventilation; End of life; Extubation; Terminal weaning; Complicated grief
MeSH Terms: conditions — Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Withdrawal of mechanical ventilation

SUMMARY:
The purpose of the study is to assess the dying process in critically ill patients with decision to withdraw invasive mechanical ventilation in anticipation of death and to compare effects of extubation and those of terminal weaning of mechanical ventilation on relatives and care givers. The investigators primary hypothesis is that extubation is associated with less symptoms of post-traumatic stress disorders in relatives, as compared to terminal weaning.

ELIGIBILITY:
Inclusion Criteria:

* End of life decision to withdraw invasive mechanical ventilation after at least 48 hours of ICU stay

Exclusion Criteria:

* Age under 18 years
* Non invasive mechanical ventilation
* Brain death
* Death before withdrawal of mechanical ventilation
* No French-speaking relative
* Refusal of relative to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in ICU with end of life decision to withdraw invasive mechanical ventilation after at least 48 hours of ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Post traumatic Stress Disorder | three month after patient's death
  Post traumatic Stress Disorder as assessed by the Impact of event Scale-revised(IES-R)

SECONDARY OUTCOMES:
Post traumatic Stress Disorder | 12 months after patient's death
  Post traumatic stress disorder of relatives assessed by the Impact of Event Scale -revised (IES-R)
Anxiety and depression | 3, 6 and 12 months after patient's death
  Anxiety and depression of the relatives, assessed by the hospital Anxiety and Depression Scale (HADS)
Complicated grief | 6 and 12 months after patient's death
  Complicated grief as assessed by the Inventory of Complicated Grief (ICG) scale
Relative's satisfaction | 3 months after patient's death
  Questionnaire on relative's satisfaction
Nurse's satisfaction | within day 1 after patient's death
  Questionnaire on nurse's satisfaction
Physician's satisfaction | within day 1 after patient's death
  Questionnaire on physician's satisfaction
Burn out syndrome of the nurse | within day 1 after patient's death
  Burn out syndrome of the patient's nurse as assessed by the Job Strain scale
Burn out syndrome of the physician | within day 1 after patient's death
  Burn out syndrome of the patient's physician as assessed by the Job Strain scale

CONTACTS AND LOCATIONS:
Overall Officials: Jean Reignier, MD, PhD, Principal Investigator — Centre Hospitalier Départemental de la Vendée, La Roche sur Yon, France; René Robert, MD, Principal Investigator — Poitiers University Hospital
Locations (44):
- France (44):
  - Réanimation médicale CHU, Angers
  - Réanimation, CH d'Angoulême, Angoulême
  - Réanimation, CH d'Annecy, Annecy
  - Réanimation, Belfort
  - CHU Pellegrin Tripode, Bordeaux
  - Réanimation, CHU, Bordeaux
  - CHU Ambroise Paré, Boulogne
  - CHU La Cavale Blanche, Brest
  - CHU de Côte de Lumière, Caen
  - Centre Hospitalier, Service de réanimation, Charleville-Mézières
  - CH de Chartres, Chartres
  - CHU Gabriel Montpied, Clermont Ferrand, Clermont-Ferrand
  - CHU Louis Mourier, Colombes
  - CH de Dieppe, Dieppe
  - CHU Dijon, Dijon
  - CHU Raymond Poincaré, Garches
  - CHU Grenoble, Grenoble
  - CHD de la Vendée, La Roche-sur-Yon
  - CH de La Rochelle, La Rochelle
  - CH du Mans, Le Mans
  - CH du Puy, Le Puy-en-Velay
  - CH Docteur Schaffner, Lens
  - CHU de Lille, Lille
  - CH de Lorient, Lorient
  - CHU Marseille, Hopital La Timone, Marseille
  - CHU de Marseille, Hopital Nord, Marseille
  - CH Marc Jacquet, Melun
  - CH de Montauban, Montauban
  - CHI André Grégoire, Montreuil
  - CH de Mulhouse, Mulhouse
  - CHU de Nantes - Hôtel Dieu, Nantes
  - CHU Orléans - Réanimation Médicale, Orléans
  - CHU Saint Louis, Paris
  - CHU Paris Cochin, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - CHU Hopital Européen Georges Pompidou, Paris
  - CHU Lariboisière, Paris
  - CHU Poitiers, Poitiers
  - CH de Roanne, Roanne
  - Hôpital Delafontaine, Saint-Denis
  - CH de Saint-Nazaire, Saint-Nazaire
  - Hôpital Foch, Suresnes
  - CHU Tours, Tours
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Robert R, Le Gouge A, Kentish-Barnes N, Cottereau A, Giraudeau B, Adda M, Annane D, Audibert J, Barbier F, Bardou P, Bourcier S, Bourenne J, Boyer A, Brenas F, Das V, Desachy A, Devaquet J, Feissel M, Ganster F, Garrouste-Orgeas M, Grillet G, Guisset O, Hamidfar-Roy R, Hyacinthe AC, Jochmans S, Jourdain M, Lautrette A, Lerolle N, Lesieur O, Lion F, Mateu P, Megarbane B, Merceron S, Mercier E, Messika J, Morin-Longuet P, Philippon-Jouve B, Quenot JP, Renault A, Repesse X, Rigaud JP, Robin S, Roquilly A, Seguin A, Thevenin D, Tirot P, Vinatier I, Azoulay E, Reignier J. Terminal weaning or immediate extubation for withdrawing mechanical ventilation in critically ill patients (the ARREVE observational study). Intensive Care Med. 2017 Dec;43(12):1793-1807. doi: 10.1007/s00134-017-4891-0. Epub 2017 Sep 22. PMID 28936597